CLINICAL TRIAL: NCT01714089
Title: A Phase II Study Evaluating RNS60 Compared to Interferon Beta-1a (Avonex) for the Treatment of Relapsing Remitting Multiple Sclerosis
Brief Title: Proof of Concept Study Evaluating RNS60 in the Treatment of Relapsing Remitting Multiple Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06.1.1.H1
Record Dates: First submitted 2012-10-19; First posted 2012-10-25 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Relapsing remitting multiple sclerosis; RR-MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — RNS60; Interferon beta-1a

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- RNS60 125 ml (Experimental): 125 ml of RNS60 administered weekly by IV infusion
  Interventions: Drug: RNS60 125 ml
- RNS60 250 ml (Experimental): 250 ml of RNS60 administered weekly by IV infusion
  Interventions: Drug: RNS60 250 ml
- Interferon beta-1a (Active Comparator): Weekly dose of 30 mcg Interferon beta-1a (Avonex) administered by intramuscular injection.
  Interventions: Drug: Interferon beta 1a

INTERVENTIONS:
Drug: RNS60 125 ml
  Arms: RNS60 125 ml
Drug: RNS60 250 ml
  Arms: RNS60 250 ml
Drug: Interferon beta 1a
  Arms: Interferon beta-1a

SUMMARY:
The purpose of this study is to determine whether RNS60 is effective in the treatment of RR-MS compared to interferon beta-1a.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged between 18 and 50 years.
2. Diagnosis of RR-MS according to McDonald 2010 diagnostic criteria with a prior brain MRI that demonstrates lesions consistent with RRMS, both within the past year.
3. No evidence of relapse during the 60 days prior to enrollment.
4. EDSS score of 0-5 at screening.
5. Women of childbearing potential who have a negative pregnancy test (serum HCG) at screening.
6. Men or women of reproductive potential who commit to use adequate contraception during the study and for 1 month following the last day of treatment.
7. Subjects must be capable of understanding the purpose and risks of the study and provide written, informed consent.

Exclusion Criteria:

1. Diagnosis of Secondary Progressive MS, Primary Progressive MS or Progressive Relapsing MS.
2. Normal baseline brain MRI.
3. History of any clinically significant autoimmune disease: inflammatory bowel disease, diabetes, lupus or severe asthma.
4. Current or prior malignancies (excluding non-melanoma skin carcinoma or in situ carcinoma of the cervix that has been adequately treated.)
5. Significant organ dysfunction, including cardiac, renal (eGFR ≤ 60 ml/min.), liver, central nervous system, pulmonary, vascular, gastrointestinal, endocrine, or metabolic (e.g., creatinine ≥ 1.6 mg/dL; ALT or AST ≥ 1.5x the upper limit of normal), history of myocardial infarction, congestive heart failure, or arrhythmias within 6 months prior to enrollment.
6. Steroid therapy within 60 days prior to enrollment, with the exception of corticosteroids or ACTH for relapse treatment during the course of the study.
7. Known allergy to Gadolinium-DTPA
8. Therapy with any immunomodulatory drugs within 3 months prior to enrollment, including but not limited to interferons, glatiramir acetate, BG-12, teriflunomide, laquinimod and IV immunoglobulin.
9. Treatment at any time with immunosuppressive drugs such as cladribine, total lymphoid irradiation, monoclonal antibody treatment, mitoxantrone, Tysabri, fingolimod, cytoxan, methotrexate.
10. Participation in any investigational therapy within one year prior to enrollment, unless given approval by PI.
11. Known or suspected current or past alcohol or drug abuse within one year prior to enrollment.
12. Any medical, psychiatric or other condition that could result in a subject not being able to comply with protocol requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in number of GAD-enhancing lesions from baseline | 3, 4, 5, and 6 months
  Cumulative number of GAD-enhancing lesions by MRI at months 3, 4, 5, and 6

SECONDARY OUTCOMES:
Change in number of T2 lesions from baseline | Months 3, 4, 5, and 6
  Cumulative number of new or newly enlarged T2 lesions over 6 months of treatment
Brain volume | 6 months
  Brain volume by MRI over 6 months of treatment
T2 lesion volume | 6 month
  T2 lesion volume by MRI over 6 months of treatment
Annualized Relapse Rate | 6 months
  Annualized Relapse Rate over 6 months
Expanded Disability Status Scale (EDSS), change from baseline | 3, 6 months
  Progression of disability as assessed by the Expanded Disability Status Scale at months 3 and 6.
Multiple Sclerosis Functional Composite, change from baseline | 3, 6 months
  Progression of disability as assessed by the Multiple Sclerosis Functional Composite tool at months 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Lublin, MD, PhD, Principal Investigator — Mt. Sinai School of Medicine
Locations (1):
- Mt. Sinai School of Medicine, New York, New York, United States